CLINICAL TRIAL: NCT00413946
Title: Neuroprotective Effect of High Dose Erythropoietin in Very Preterm Infants
Brief Title: Does Erythropoietin Improve Outcome in Very Preterm Infants?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Neonatal Network (Network)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Bucher Hans Ulrich, full professor of Neonatology, Swiss Neonatal Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3200B0-108176; RoFAR ID 2127989593 (Other Grant/Funding Number: 3200B0-108176); 3200B0-108176 (Other Grant/Funding Number: SNF 3200B0-108176)
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Intracranial Hemorrhage; Periventricular Leukomalacia; Cerebral Palsy; Developmental Psychomotor Disorders
Keywords: Premature infant; developmental outcome
MeSH Terms: conditions — Intracranial Hemorrhages; Leukomalacia, Periventricular; Cerebral Palsy; Psychomotor Disorders; Premature Birth | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental): Three doses of rErythropoietin (3000 U/kg body weight) intravenously at 3, 12-18 and 36-42 hours after birth.
  Interventions: Drug: Recombinant human Erythropoietin
- saline (Placebo Comparator): Three doses of placebo (0.9% saline 1 ml/kg body weight) intravenously at 3, 12-18 and 36-42 hours after birth
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Recombinant human Erythropoietin — 3 doses 3000 units (1 ml) of recombinant human erythropoietin per kg body weight
  Arms: Erythropoietin
Drug: saline — three doses of 1.0 ml saline per body weight
  Other Names: NaCl 0.9%
  Arms: saline

SUMMARY:
The main goal of this trial is to investigate whether early administration of human erythropoietin (EPO) in very preterm infants improves neurodevelopmental outcome at 24 months corrected age.

This study is designed as randomized, double-masked, placebo controlled multicenter study involving at least 420 patients.

DETAILED DESCRIPTION:
HYPOTHESIS Early administration of human erythropoietin (EPO) in very preterm infants reduces perinatal injury to the brain (retina), lung and gut and improves neurodevelopmental outcome at 24 months corrected age.

PRIMARY OBJECTIVE To determine whether cerebral outcome is improved if infants born between 26 0/7 and 31 6/7 gestational weeks at birth receive erythropoietin in high dose in the first three days after birth.

SECONDARY OBJECTIVES To determine whether early administration of EPO alters the incidence of complications typically associated with preterm birth, i.e. mortality, septicaemia, necrotising enterocolitis, bronchopulmonary dysplasia (oxygen dependency at 36 weeks postmenstrual age), retinopathy, intracranial haemorrhage, white matter disease (periventricular leucomalacia), growth failure, cerebral palsy and handicap at 5 years.

Biomarkers of encephalopathy of prematurity assessed on magnetic resonance imaging (MRI) at term equivalent age.

RATIONALE EPO has been shown to be protective against hypoxic-ischaemic and inflammatory injuries in a broad range of tissues and organs besides promoting red cell formation. It has been shown to have neuroprotective and neurotrophic activity in animals after acute brain damage as well as in adult stroke patients. Several mechanisms explaining this activity have been recognized: EPO inhibits glutamate release in the brain, modulates intracellular calcium metabolism, induces the generation of anti-apoptotic factors, reduces inflammation, decreases nitric oxide-mediated injury, and has direct antioxidant effects.

Very preterm infants have significant delay in mental and physical development assessed at 24 months corrected age. The most critical period are the first days after preterm birth where the oxygenation of the brain may be impaired by respiratory, circulatory and nutritional insufficiency. Although there are probably several mechanisms involved in permanent brain damage, it is most likely that EPO with its multiple action may reduce this damage.

EPO has been studied in several trials in preterm infants to prevent anaemia and is now widely used for this indication.

STUDY DESIGN Randomized, double-masked, placebo-controlled multicenter clinical trial. Research plan 420 infants will be randomized during the first three hours of life to receive EPO (3000 U/kg body weight) or placebo intravenously at 3, 12-18 and 36-42 hours after birth. Standardized evaluation including cerebral sonography at day 1 and 7 and at 36 0/7 gestational weeks (or at discharge home if discharged before) will determine the presence or absence of complications. Cerebral volume and white matter volume will be assessed at 40 postmenstrual weeks with MRI (only if available).

Experienced examiners will assess developmental function at 24 months corrected age using the reliable and validly revised Bayley Scales II of Infant Development and determine the presence or absence of impairment of motor function (cerebral palsy) and neurosensory function (blindness or deafness).

CLINICAL SIGNIFICANCE At least 1 of every 100 live born infants is born very preterm. 90% of these infants survive but >50% have a delay in mental and physical development assessed at 24 months corrected age. More subtle problems affecting cognition, vision and hearing are common at the age of five years and have an impact on school performance and quality of life of the infants and their families. The aim of this trial is to examine whether a short, easily applicable and well tolerated pharmacological intervention can improve neurodevelopmental outcome.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 26 0/7 and 31 6/7 gestational weeks
* Postnatal age less than 3 hours
* Informed parental consent (preferably obtained before birth)

Exclusion Criteria:

* Genetically defined syndrome
* Severe congenital malformation adversely affecting life expectancy
* Severe congenital malformation adversely affecting neurodevelopment
* A priory palliative care
* Intracranial haemorrhage grade 3 or more detected before dose 3 of Erythropoietin

Max Age: 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mental developmental index (Bayley II) and motor, visual and hearing impairment | at age of 24 months corrected for prematurity.

SECONDARY OUTCOMES:
MRI at term equivalent | 40 postmenstrual weeks
  White matter injury score grey matter injury score brain maturation
cerebral palsy. | First 24 months of life (corrected for prematurity)
Cognitive development and cerebral palsy | 5 years
  Kaufmann ABC II, standardized neurological, visual and hearing examination, questionnaire about health status and behavior.
  Classification of impairments, disabilities and handicaps.

CONTACTS AND LOCATIONS:
Overall Officials: Hans U Bucher, Prof, Principal Investigator — University of Zurich
Locations (5):
- Switzerland (5):
  - Kantonsspital, Aarau
  - Kantonsspital, Basel
  - Kantonsspital, Chur
  - Hopital universitaire, Geneva
  - University Hospital, Zurich

REFERENCES:
- [Result] Fauchere JC, Dame C, Vonthein R, Koller B, Arri S, Wolf M, Bucher HU. An approach to using recombinant erythropoietin for neuroprotection in very preterm infants. Pediatrics. 2008 Aug;122(2):375-82. doi: 10.1542/peds.2007-2591. PMID 18676556
- [Derived] Picotti E, Reinelt T, Koller B, Bucher HU, Ruegger CM, Fauchere JC, Natalucci G; Swiss EPO Neuroprotection Trial Group. Effect of Early High-Dose Recombinant Human Erythropoietin on Behavior and Quality of Life in Children Aged 5 Years Born Very Preterm: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2245499. doi: 10.1001/jamanetworkopen.2022.45499. PMID 36477478
- [Derived] Natalucci G, Latal B, Koller B, Ruegger C, Sick B, Held L, Bucher HU, Fauchere JC; Swiss EPO Neuroprotection Trial Group. Effect of Early Prophylactic High-Dose Recombinant Human Erythropoietin in Very Preterm Infants on Neurodevelopmental Outcome at 2 Years: A Randomized Clinical Trial. JAMA. 2016 May 17;315(19):2079-85. doi: 10.1001/jama.2016.5504. PMID 27187300
- [Derived] Fauchere JC, Koller BM, Tschopp A, Dame C, Ruegger C, Bucher HU; Swiss Erythropoietin Neuroprotection Trial Group. Safety of Early High-Dose Recombinant Erythropoietin for Neuroprotection in Very Preterm Infants. J Pediatr. 2015 Jul;167(1):52-7.e1-3. doi: 10.1016/j.jpeds.2015.02.052. Epub 2015 Apr 8. PMID 25863661
- [Derived] O'Gorman RL, Bucher HU, Held U, Koller BM, Huppi PS, Hagmann CF; Swiss EPO Neuroprotection Trial Group. Tract-based spatial statistics to assess the neuroprotective effect of early erythropoietin on white matter development in preterm infants. Brain. 2015 Feb;138(Pt 2):388-97. doi: 10.1093/brain/awu363. Epub 2014 Dec 22. PMID 25534356
- [Derived] Leuchter RH, Gui L, Poncet A, Hagmann C, Lodygensky GA, Martin E, Koller B, Darque A, Bucher HU, Huppi PS. Association between early administration of high-dose erythropoietin in preterm infants and brain MRI abnormality at term-equivalent age. JAMA. 2014 Aug 27;312(8):817-24. doi: 10.1001/jama.2014.9645. PMID 25157725
- [Derived] Ruegger CM, Kraus A, Koller B, Natalucci G, Latal B, Waldesbuhl E, Fauchere JC, Held L, Bucher HU. Randomized controlled trials in very preterm infants: does inclusion in the study result in any long-term benefit? Neonatology. 2014;106(2):114-9. doi: 10.1159/000362784. Epub 2014 Jun 20. PMID 24969309
- [Derived] Dame C, Langer J, Koller BM, Fauchere JC, Bucher HU. Urinary erythropoietin concentrations after early short-term infusion of high-dose recombinant epo for neuroprotection in preterm neonates. Neonatology. 2012;102(3):172-7. doi: 10.1159/000339283. Epub 2012 Jul 4. PMID 22776958
- See also: Swiss Neonatal Network — http://www.neonet.ch